CLINICAL TRIAL: NCT05988255
Title: Efficacy of Static Progressive Stretching Technique Versus Traditional Stretching in Primary Adhesive Capsulitis: a Randomized Controlled Trial
Brief Title: Efficacy of Static Progressive Stretch Versus Traditional Stretch in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Ramadan Ibrahim Abdul-ghani El Deab, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004172
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Adhesive Capsulitis; Stretch; Physical Neglect
Keywords: Adhesive capsulitis; Static progressive stretch
MeSH Terms: conditions — Bursitis | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Prospective single-blinded randomized controlled trial (therapy, level 1B)
Who Masked: Participant
Masking Description: Participants were blinded to which treatment they would receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static progressive stretch (Experimental)
  Interventions: Device: Static progressive stretching
- Cyclic manual stretch (Active Comparator)
  Interventions: Other: Cyclic manual stretching
- No treatment (No Intervention)

INTERVENTIONS:
Device: Static progressive stretching — A stretching technique applies a mechanical progressive stretch
  Other Names: Stretching exercises
  Arms: Static progressive stretch
Other: Cyclic manual stretching — A stretching technique applies an intermittent manual stretch
  Other Names: Stretching exercises
  Arms: Cyclic manual stretch

SUMMARY:
This study will be conducted to compare the effectiveness of static progressive stretching using the joint active system (JAS) shoulder device with cyclic manual stretching and controls on shoulder range of motion (ROM), time to gain ROM, and function in patients with adhesive capsulitis. The study includes three groups. Group A (15 patients) will receive static progressive stretch using the JAS device. Group B (15 patients) will receive cyclic manual stretching in flexion, abduction, and external and internal rotations. Group C (15 patients) is a control group that will receive no treatment until the end of the study.

DETAILED DESCRIPTION:
The study design: Prospective single-blinded randomized controlled trial (therapy, level 1B). A flow diagram according to the Consolidated Standards of Reporting Trials (CONSORT) statement will be presented to illustrate the progression of the study.

The sample size is calculated using G*power software (version 3.1.9.7, Franz Faul, Universitat Kiel, Germany) and it suggests that 42 participants (14 per group) will be needed using the MANOVA test. Cohen's d is set to be 0.25 with 80% power (alpha = 0.05) to detect an effect size.

Patients are randomly assigned to either of three groups (A, B, or C) using a computer-generated list. They are allocated by an outside party who isn't involved in the treatment using sequentially numbered sealed envelopes.

Inclusion criteria: (1) Patients of both genders with unilateral primary adhesive capsulitis (2) Patients aged between 40-65. (3) Pain duration of three months or more. (4) Range of motion loss of greater than 25% in at least 2 planes and passive external rotation loss that is greater than 50% of the uninvolved shoulder or less than 30° of external rotation.

Exclusion criteria: (1) Previous surgery or manipulation under anesthesia. (2) Other conditions affecting the shoulder as (rheumatoid arthritis, osteoarthritis, rotator cuff disease, or malignancies). (3) Neurological deficits affecting shoulder function.

Demographic data will be collected for all subjects regarding age, gender, dominance, and painful side. After patient selection according to the inclusion and exclusion criteria, we will measure shoulder range of motion (ROM) using a Baseline Digital Absolute Axis Goniometer, and shoulder function using the SPADI scale.

Range of motion will be assessed at baseline (before the start of treatment), at the end of each week, and at the end of 12 weeks.

Shoulder function will be assessed using SPADI at baseline (before the start of treatment) and at the end of treatment.

The mean time needed to reach ROM at 3 months will be assessed in each group and compared between groups.

Treatment procedures:

All patients in the three groups will be educated about the natural history of the disease and instructed to stay active at home through encouraging activity modification without pain. Each patient in the treatment groups will receive two treatment sessions per week for a series of 12 weeks.

1. Static progressive stretching using JAS shoulder device (Group A): The static progressive stretch device applies stretch toward external and internal rotation from different degrees of scapular plane abduction. After adjustment of the device, it will be worn for 45 minutes (30 minutes stretching toward external rotation and 15 minutes toward internal rotation). The stretch position will be held for a series of 5 minutes and rest in between according to patient tolerance.
2. Cyclic manual stretching (Group B): Five to twenty seconds of stretching and 10 seconds of rest will be used 10 times in each of the following directions (flexion, scapular plane abduction, external rotation, and internal rotation) and stretch to target rotator cuff interval. The stretching dose will be determined based on the patient's level of irritability.
3. Group C: Fifteen patients will receive no physiotherapy treatment until the end of the study. As an ethical consideration, subjects in this group will receive the full treatment after the end of the study after data collection.

Statistical analysis:

Data will be analyzed using the statistical package for social sciences (SPSS) computer program version 24 software (IBM SPSS Inc., Chicago, IL, USA).

Descriptive statistics will be expressed as mean ± standard deviation for continuous variables.

The normality of data will be examined using Kolmogorov-Smirnov statistical test.

Repeated measures ANOVA test will be used to determine the difference between baseline and post-treatment scores for the ROM and time to gain ROM within each group.

Wilcoxon signed-rank test will be used to determine the difference between baseline and post-treatment scores for pain and function.

Kruskal Wallis ANOVA will be used for pain and function scores difference between groups (ordinal data).

A MANOVA test will be used to identify the difference between the three groups regarding ROM (flexion, extension, abduction, internal rotation, external rotation in adduction, and external rotation in abduction).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with unilateral primary adhesive capsulitis.
2. Patients aged between 40-65.
3. Pain duration of three months or more.
4. Range of motion loss of greater than 25% in at least 2 planes and passive external rotation loss that is greater than 50% of the uninvolved shoulder or less than 30° of external rotation.

Exclusion Criteria:

1. Previous surgery or manipulation under anesthesia.
2. Other conditions affecting the shoulder as (rheumatoid arthritis, osteoarthritis, rotator cuff disease, or malignancies).
3. Neurological deficits affecting shoulder function.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Range of motion | Three months
  Shoulder flexion, extension, abduction, external rotation and internal rotation will be measured using Baseline Digital Absolute Axis Goniometer
Function | Three months
  The patient will be advised to select the number that best reflects the intensity of their discomfort and the degree of trouble they are having using the affected shoulder using SPADI.

SECONDARY OUTCOMES:
Time to gain range motion | Three months
  Mean time needed to reach ROM at 3 months will be assessed in each group and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided